CLINICAL TRIAL: NCT01681628
Title: Effectiveness of Thought Field Therapy Provided by Newly Instructed Community Workers to a Traumatized Population in Uganda: A Randomised Trial
Brief Title: Community Self-help Using Thought Field Therapy in a Traumatised Population in Uganda: a Randomised Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thought Field Therapy Foundation (UK) Ltd (Other)
Collaborators: Thought Field Therapy Foundation. (Unknown); Mats Uldal Humanitarian Foundation (Unknown)
Responsible Party: Principal Investigator, Robert Howard Robson, Dr Robert Howard Robson, Thought Field Therapy Foundation (UK) Ltd
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Uganda2012
Record Dates: First submitted 2012-09-02; First posted 2012-09-10 (Estimated); Results first posted 2017-05-01 (Actual); Last update posted 2017-05-01 (Actual); Status verified 2017-03

CONDITIONS: Post-traumatic Stress Disorder
Keywords: Thought Field Therapy.; Post-traumatic stress disorder.; Post-traumatic stress disorder check list for Civilians.; Uganda; Ugandan therapists.; Community treatment.
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thought Field Therapy (Experimental): Thought Field Therapy delivered by trained community leaders.
  Interventions: Behavioral: Thought Field Therapy.
- Wait list (Other): Delayed intervention.
  No intervention prior to assessment after one week (pre-test 2). Then treated with Thought Field Therapy, and re-assessed after a further week (post-test).
  Interventions: Behavioral: Thought Field Therapy.

INTERVENTIONS:
Behavioral: Thought Field Therapy. — Thought Field Therapy is a meridian based therapy, where clients tap on specific parts of their body, according to a particular protocol. This does not obliterate the memory of the trauma, but relieves the associated distress.

SUMMARY:
Thought Field Therapy (TFT) is a simple technique that involves tapping on points of the body corresponding to the meridians used in acupuncture. By using specific sequences, TFT can be used to treat a variety of psychological problems. Patients can be taught to treat themselves, and lay people can be trained to treat others in their community, as has been shown for narrative exposure therapy.

Thought Field Therapy has been used to treat whole communities who have suffered psychological trauma following natural disasters and violent conflicts. In these circumstances, TFT can be used as a stand-alone therapy, or as an adjunct to other psychological therapies, by removing the pain of re-living the traumatic events.

Studies in Rwanda have shown that individuals within a community can be treated with brief TFT sessions. Both short-term and longer-term improvements in scores of Post-Traumatic Stress Disorder (PTSD) measurement scales have been demonstrated.

The Kasese District in Uganda has suffered from factional conflicts and the consequences of the ongoing struggles in neighbouring countries for many years. Although the government has controlled the situation and secured the borders, many are still haunted by the psychological consequences.

The purpose of the study is to validate the model of addressing widespread psychological trauma following conflict by training community leaders to help others in their community using TFT.

Thirty-six community leaders will be given a two-day training in algorithm level trauma-relief TFT. They will then treat 128 volunteers for their traumas, using TFT, who will be assessed before and one week after treatment by the post-traumatic stress disorder check-list questionnaire for civilians (PCL-C). As a control, a further 128 volunteers will join a wait-list group, who will be assessed at the same time, but treated later.

PCL-C scores before and after treatment will be compared with the wait-list group scores before and after waiting, but before their treatment.

A follow-up assessment of the participants will be undertaken 1 to 2 years later.

DETAILED DESCRIPTION:
Six TFT practitioners from the USA, Great Britain, and Norway will train 36 community leaders during a two-day trauma-relief training programme. These newly-trained practitioners will then treat 256 volunteers who feel that they are suffering from psychological trauma. The six visiting practitioners, together with two additional TFT practitioners from Rwanda, will supervise and support the study following the training.

A Catholic Priest, Father Peter Mubunga Basaliza, on behalf of the Kasese Diocese, will organise the recruitment of the local trainers and volunteer participants, including publicising by local radio. All faiths will be welcome, but volunteers must be 18 years of age or older. Volunteers will be informed of their allocated date and time to attend for inclusion in the study. Any volunteer who cannot be accommodated in the study because the pre-requisite number has been met, will be offered TFT by the visiting practitioners and trained community leaders.

Signed consent will be obtained prior to commencing the study. Participants will be provided with an information sheet and duplicate consent forms in Lhukonzo (the local language), and assistance will be provided by Ugandan therapists for those who have difficulty reading. Consent forms will also be available in English for those for whom it is the preferred language. Each participant will also complete a demographic questionnaire.

Participants will be free to withdraw at any time, and any who do so will still be offered TFT, if desired.

Sixty-four participants will be seen each day, 32 in the morning, and 32 in the afternoon, for four consecutive days. They will be allocated according to a previously computer generated random number sequence, to Group A and provided with a blue folder, or Group B and provided with a red folder. Their names will be recorded on a sign-in sheet. They will be identified by a number, which will be written on their folder and documents. Both groups will initially complete the post-trauma checklist (PCL-C) questionnaire (www.pdhealth.mil) available in Lhukonzo, referring to symptoms within the previous week. Therapists, who will be unaware of the individual's group allocation, will assist if necessary. The PCL-C has been translated from English into Lhukonzo and back into English to ensure that the translation is accurate.

The PCL-C consists of 17 questions, each question scoring from 1 - 5. Thus the minimum score is 17 and maximum score 85. A score of 17 has no features of PTSD and 85 the highest score for PTSD. When used as a screening tool, a score of more than 50 is considered to be diagnostic of PTSD.

Completed questionnaires and consent forms will be kept in their folders and retained by the researchers.

Following completion of their PCL-C forms, Group A participants will be treated using Thought Field Therapy by the newly trained therapists for their traumas, supervised by the researchers. The therapists will keep a record for each participant of the problem that was treated, algorithms used, the time taken, and the Subjective Units of Distress (SUD) scores (0-10).

Group B will be a control (wait-list group) and will receive no treatment following their first visit. This model has been successfully utilised in Rwanda.

One week later, at the same time and day of the week as they first attended, the participants in group A and group B will return and repeat their PCL. On this occasion, testing will be followed by treatment for Group B.

After a further week, Group B only will return for repeat testing using PCL.

In summary, the protocol to be followed will be:

* Two-day training of new therapists
* Day one of study: 9am - PCL test of 16 Group A and 16 Group B 11am -Treat the 16 Group A

  1pm - Test a new group of 16 A and 16 B 3pm - Treat the new 16 group A
* Days 2-4: Same as for day one, but with new participants. Each therapist will treat the same number in each group.
* Days 8-11 9am -PCL test of 16 Group A and 16 Group B 11am -Treat the 16 Group B

  1pm - Test another 16 of each Group 3pm -Treat the new Group B
* Day 18 Test all Group B, 16 every two hours from 9am

Mean + SD PCL test scores will be calculated for each group during their four days of each week, and of Group B on day 18. That is:

Group A days 1-4 (A pre-treatment) Group B days 1-4 (B pre-treatment) Group A days 8-11 (A post-treatment) Group B days 8-11 (B post-no treatment) Group B day 18 (B post-treatment)

The statistical significance of differences of mean scores will be analysed by analysis of variance and paired samples t tests. Significances of differences in group proportions with diagnostic scores for PTSD will be assessed by a non-parametric test.

Statistically significant differences were found in a similar study in Rwanda, with smaller numbers, so the study will be adequately powered.

A follow-up assessment will be done 19 months later.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers recruited from local communities, who feel that they are suffering from psychological trauma.

Exclusion Criteria:

* Minimum age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2012-06; Primary Completion 2012-07 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert H Robson, MA MB BChir, Principal Investigator — Thought Field Therapy Foundation (UK) Ltd
Locations (1):
- St Augustine's Catechist Training Centre, PO Box 155, Kasese, Kasese, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Spreadsheet available on request. Individual paper copies also available.

REFERENCES:
- [Background] Callahan RJ. Tapping the healer within. New York, NY: McGraw-Hill, 2001
- [Background] Connolly S, Sakai C. Brief trauma intervention with Rwandan genocide-survivors using thought field therapy. Int J Emerg Ment Health. 2011;13(3):161-72. PMID 22708146
- [Background] Ertl V, Pfeiffer A, Schauer E, Elbert T, Neuner F. Community-implemented trauma therapy for former child soldiers in Northern Uganda: a randomized controlled trial. JAMA. 2011 Aug 3;306(5):503-12. doi: 10.1001/jama.2011.1060. PMID 21813428
- [Background] Feinstein D. Energy psychology in disaster relief. Traumatology 14: 127-129, 2008.
- [Background] Sakai CE, Connolly SM, Oas P. Treatment of PTSD in Rwandan child genocide survivors using thought field therapy. Int J Emerg Ment Health. 2010 Winter;12(1):41-9. PMID 20828089
- [Background] Bisson JI, Roberts NP, Andrew M, Cooper R, Lewis C. Psychological therapies for chronic post-traumatic stress disorder (PTSD) in adults. Cochrane Database Syst Rev. 2013 Dec 13;2013(12):CD003388. doi: 10.1002/14651858.CD003388.pub4. PMID 24338345
- [Background] Blanchard EB, Jones-Alexander J, Buckley TC, Forneris CA. Psychometric properties of the PTSD Checklist (PCL). Behav Res Ther. 1996 Aug;34(8):669-73. doi: 10.1016/0005-7967(96)00033-2. PMID 8870294
- [Background] Church D, Hawk C, Brooks AJ, Toukolehto O, Wren M, Dinter I, Stein P. Psychological trauma symptom improvement in veterans using emotional freedom techniques: a randomized controlled trial. J Nerv Ment Dis. 2013 Feb;201(2):153-60. doi: 10.1097/NMD.0b013e31827f6351. PMID 23364126
- [Background] Church D, Yount G, Brooks AJ. The effect of emotional freedom techniques on stress biochemistry: a randomized controlled trial. J Nerv Ment Dis. 2012 Oct;200(10):891-6. doi: 10.1097/NMD.0b013e31826b9fc1. PMID 22986277
- [Background] Connolly SM, Roe-Sepowitz D, Sakai C, Edwards J. Utilizing community resources to treat PTSD: randomised controlled study using thought field therapy. African Journal of Traumatic Stress 3: 82-90, 2013.
- [Background] Feinstein D. Rapid treatment of PTSD: why psychological exposure with acupoint tapping may be effective. Psychotherapy (Chic). 2010 Sep;47(3):385-402. doi: 10.1037/a0021171. PMID 22402094
- [Background] Feinstein D. Acupoint stimulation in treating psychological disorders. Review of general Psychology 16: 364-380, 2012. doi: 10.1037/a0021171
- [Background] Folkes CE. Thought field therapy and trauma recovery. Int J Emerg Ment Health. 2002 Spring;4(2):99-103. PMID 12166020
- [Background] Galea S, Nandi A, Vlahov D. The epidemiology of post-traumatic stress disorder after disasters. Epidemiol Rev. 2005;27:78-91. doi: 10.1093/epirev/mxi003. No abstract available. PMID 15958429
- [Background] Hui KK, Liu J, Makris N, Gollub RL, Chen AJ, Moore CI, Kennedy DN, Rosen BR, Kwong KK. Acupuncture modulates the limbic system and subcortical gray structures of the human brain: evidence from fMRI studies in normal subjects. Hum Brain Mapp. 2000;9(1):13-25. doi: 10.1002/(sici)1097-0193(2000)9:13.0.co;2-f. PMID 10643726
- [Background] Jonas DE, Cusack K, Forneris CA, Wilkins TM, Sonis J, Middleton JC, Feltner C, Meredith D, Cavanaugh J, Brownley KA, Olmsted KR, Greenblatt A, Weil A, Gaynes BN. Psychological and Pharmacological Treatments for Adults With Posttraumatic Stress Disorder (PTSD) [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2013 Apr. Report No.: 13-EHC011-EF. Available from http://www.ncbi.nlm.nih.gov/books/NBK137702/ PMID 23658937
- [Background] Kim YD, Heo I, Shin BC, Crawford C, Kang HW, Lim JH. Acupuncture for posttraumatic stress disorder: a systematic review of randomized controlled trials and prospective clinical trials. Evid Based Complement Alternat Med. 2013;2013:615857. doi: 10.1155/2013/615857. Epub 2013 Feb 6. PMID 23476697
- [Background] Metcalf O, Varker T, Forbes D, Phelps A, Dell L, DiBattista A, Ralph N, O'Donnell M. Efficacy of Fifteen Emerging Interventions for the Treatment of Posttraumatic Stress Disorder: A Systematic Review. J Trauma Stress. 2016 Feb;29(1):88-92. doi: 10.1002/jts.22070. Epub 2016 Jan 7. PMID 26749196
- [Background] Reed RV, Fazel M, Goldring L. Post-traumatic stress disorder. BMJ. 2012 Jun 25;344:e3790. doi: 10.1136/bmj.e3790. No abstract available. PMID 22734075
- [Background] Stone B, Leyden L, Fellows B. Energy Psychology treatment for post traumatic stress in genocide survivors in a Rwandan orphanage: a pilot investigation. Energy Psychology 1: 73-81, 2009.
- [Background] Stone B, Leyden L, Fellows B. Energy Psychology treatment for orphan heads of households in Rwanda. Energy Psychology 2: 31-38, 2010.
- [Background] Watts BV, Schnurr PP, Mayo L, Young-Xu Y, Weeks WB, Friedman MJ. Meta-analysis of the efficacy of treatments for posttraumatic stress disorder. J Clin Psychiatry. 2013 Jun;74(6):e541-50. doi: 10.4088/JCP.12r08225. PMID 23842024
- [Result] Dunnewold AL. Thought Field Therapy efficacy following large scale traumatic events. Current Research in Psychology 5: 34-39, 2014. DOI: 10.3844/crpsp.2014.34.39
- [Result] Robson RH, Robson PM, Ludwig R, Mitabu C, Phillips C. Effectiveness of Thought Field Therapy Provided by Newly Instructed Community Workers to a Traumatized Population in Uganda: A Randomized Trial. Current Research in Psychology http://thescipub.com/PDF/ofsp.10454.pdf, 2016.
- See also: Background to local conflicts potentially causing post-traumatic stress disorder. — http://en.wikipedia.org/wiki/Rwenzururu
- See also: Co-sponsor — http://www.tftfoundation.org
- See also: Co-sponsor — http://matsuldalhumanitarianfondation.wordpress.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Public announcement throughout Kasese district of Uganda for those with symptoms of PTSD (described in announcement).
Pre-assignment Details: Participants had been previously identified. As an excess number presented, only sufficient for the trial were assigned. One participant was excluded as not meeting age criteria (had to be 18 years old or over).
Groups:
- Wait List: Delayed intervention.
  No intervention prior to assessment after one week (pre-test 2). Then treated with Thought Field Therapy, and re-assessed after a further week (post-test).
  Thought Field Therapy.: Thought Field Therapy is a meridian based therapy, where clients tap on specific parts of their body, according to a particular protocol. This does not obliterate the memory of the trauma, but relieves the associated distress.
Period: Time 1 (Entry) to Time 2 One Week Later.
Arm/Group | Thought Field Therapy | Wait List
Started | 128 | 128
Completed | 114 | 122
Not Completed | 14 | 6
Not completed — Lost to Follow-up | 14 | 6
Period: Time 2 to Time 3 (One Week Later).
Arm/Group | Thought Field Therapy | Wait List
Started | 0 (Only wait list group studied in this period.) | 122
Completed | 0 (Only wait list group studied in this period.) | 107
Not Completed | 0 | 15
Not completed — Lost to Follow-up | 0 | 15
Period: 19 Months Follow-up
Arm/Group | Thought Field Therapy | Wait List
Started | 114 | 107
Completed | 52 | 64
Not Completed | 62 | 43
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 61 | 43

BASELINE CHARACTERISTICS:
Population: Local population from Kasese district in Uganda who admitted to symptoms suggestive of PTSD and volunteered to participate. Non-attenders at Time 2 were not included in the analysis.
Groups:
- Thought Field Therapy (TFT): Thought Field Therapy delivered by trained community leaders.
  Thought Field Therapy.: Thought Field Therapy is a meridian based therapy, where clients tap on specific parts of their body, according to a particular protocol. This does not obliterate the memory of the trauma, but relieves the associated distress.
  Both groups were invited to attend 19 months later
- Wait List: Delayed intervention.
  No intervention prior to assessment after one week (pre-test 2). Then treated with Thought Field Therapy, and re-assessed after a further week (post-test).
  Thought Field Therapy.: Thought Field Therapy is a meridian based therapy, where clients tap on specific parts of their body, according to a particular protocol. This does not obliterate the memory of the trauma, but relieves the associated distress.
  Both groups were invited to attend 19 mo the later.
- Total: Total of all reporting groups
Arm/Group | Thought Field Therapy (TFT) | Wait List | Total
Number analyzed (Participants) | 114 | 122 | 236
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (16) | 45.1 (14.4) | 44.5 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 102 | 202
  Male | 14 | 20 | 34
Race/Ethnicity, Customized [Number; unit: participants]
  African (Western Uganda) | 114 | 122 | 236
PCL-C [Mean (Standard Deviation); unit: units on a scale] — PCL-C (post traumatic check list for civilians) is a measure of the severity of post traumatic stress disorder (PTSD), and can also be used for screening populations, It is a self-completed questionnaire with 17 questions scoring from 1 - 5. The scores of each question are added to create the total score for each participant. The highest possible score for any individual is 85, the lowest score being 17. A diagnostic score for PTSD is accepted as being more than 50. Participants completed the PCL-C just before treatment and one week later. The wait list group received no treatment at Time 1.
  units on a scale | 58.0 (12.6) | 61.2 (10.1) | 59.6 (11.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Post-traumatic Stress Disorder Check List for Civilians (PLC-C) Score.
Description: PCL-C (post traumatic check list for civilians) is a measure of the severity of post traumatic stress disorder (PTSD), and can also be used for screening populations, It is a self-completed questionnaire with 17 questions scoring from 1 - 5. The scores of each question are added to create the total score for each participant. The highest possible score for any individual is 85, the lowest score being 17. A diagnostic score for PTSD is accepted as being more than 50. Participants completed the PCL-C just before treatment and one week later. The wait list group received no treatment at Time 1.
  In the treatment arm, measure immediately pre-treatment (baseline) (time 1) and one week later (time 2).
  In the wait-list no therapy arm, measure at baseline (time 1), and after one week (no treatment) (time 2). The wait-list group (Thought Field Therapy group) were then treated and reassessed after a further week (time 3).
Time Frame: Baseline (Time 1), One week later (Time 2) and Two weeks later (Time 3 for Wait-list: Thought field Therapy Arm)
Population: Participants with symptoms suggestive of PTSD, excluding non-attenders at Time 2. Non-attenders at time 3 were excluded from the wait-list (Thought Field Therapy) arm.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Wait List: no Therapy: No thought field therapy intervention prior to assessment after one week (pre-test 2).
  Thought Field Therapy.: Thought Field Therapy is a meridian based therapy, where clients tap on specific parts of their body, according to a particular protocol. This does not obliterate the memory of the trauma, but relieves the associated distress.
- Wait-list: Thought Field Therapy: Received thought field therapy after second assessment (time 2) and re-assessed one week later (time 3).
  Thought Field Therapy.: Thought Field Therapy is a meridian based therapy, where clients tap on specific parts of their body, according to a particular protocol. This does not obliterate the memory of the trauma, but relieves the associated distress.
Arm/Group | Thought Field Therapy | Wait List: no Therapy | Wait-list: Thought Field Therapy
Number analyzed (Participants) | 114 | 122 | 107
units on a scale | 32.4 (14.7) | 12.4 (14.2) | 20.6 (13.5)
Statistical Analysis 1: Comparison: Thought Field Therapy vs Wait List: no Therapy; Means and differences were calculated for both groups before (time 1) and after treatment (or no treatment) (time 2). Also, the differences in mean scores from time 1 to 2 were compared between the two groups, the primary outcome. The numbers in the groups were considered adequate based on previous similar studies. The null hypothesis was that there would be no difference in any mean change in scores from time 1 to 2, between both groups; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — This was an a priori threshold; Mean Difference (Final Values) = 20.9, 95% CI 2-sided [16.1 to 24.0], Standard Error of Mean 2.0
Statistical Analysis 2: Comparison: Thought Field Therapy; Change in PCL-C scores from before to after treatment; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 32.4, 95% CI 2-sided [29.1 to 34.7], Standard Deviation 14.7
Statistical Analysis 3: Comparison: Wait List: no Therapy; Changes in PCL-C scores for control group after no treatment; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 12.4, 95% CI 2-sided [11.4 to 17.1], Standard Deviation 14.2
Statistical Analysis 4: Comparison: Wait-list: Thought Field Therapy; Change in control group PCL-C scores after treatment, that is from time 2 to time 3; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Degrees of freedom 94; Mean Difference (Final Values) = 20.6, 95% CI 2-sided [17.1 to 22.5], Standard Deviation 13.5

2. Secondary Outcome: Percentage With Scores Diagnostic for Post Traumatic Stress Disorder (PCL-C > 50) Before and After Treatment in Treatment and Control Groups.
Description: PCL-C (post traumatic check list for civilians) is a measure of the severity of post traumatic stress disorder (PTSD), and can also be used for screening populations, It is a self-completed questionnaire with 17 questions scoring from 1 - 5. The scores of each question are added to create the total score for each participant. The highest possible score for any individual is 85, the lowest score being 17. A diagnostic score for PTSD is accepted as being more than 50. Participants completed the PCL-C just before treatment and one week later. The wait list group received no treatment at Time 1.
Time Frame: Baseline (Time 1), One week later (Time 2) and Two weeks later (Time 3 for Wait-list: Thought field Therapy Arm)
Population: Participants with symptoms suggestive of PTSD, thought field therapy group treated, wait list group not treated, and wait-list group treated. All assessed one week after initial assessment and treatment, and the percentage with a score > 50 compared before and after treatment, or control.
Measure: Number; unit: percentage with PCL-C score > 50
Groups:
- Wait List no Treatment: No intervention prior to assessment after one week (pre-test 2).
  Thought Field Therapy.: Thought Field Therapy is a meridian based therapy, where clients tap on specific parts of their body, according to a particular protocol. This does not obliterate the memory of the trauma, but relieves the associated distress.
- Wait List: Thought Field Therapy: After two control assessments at times 1 and 2, the wait list group were treated and re-assessed one week later at time 3. Non-attenders at time 3 were excluded from analysis.
Arm/Group | Thought Field Therapy | Wait List no Treatment | Wait List: Thought Field Therapy
Number analyzed (Participants) | 114 | 122 | 107
percentage with PCL-C score > 50
  Time 1: number analyzed (Participants) | 114 | 122 | 0
  Time 1 | 67.5 | 82.8 |
  Time 2 | 1.8 | 41.8 | 41.8
  Time 3: number analyzed (Participants) | 0 | 0 | 107
  Time 3 |  |  | 1.9
Statistical Analysis 1: Comparison: Thought Field Therapy; Chi-squared test of any change in PCL-C from time 1 to time 2; Test type: Superiority or Other; p < 0.001, Chi-squared; percentage of participants = 65.7
Statistical Analysis 2: Comparison: Wait List no Treatment; Comparison of the percentage with diagnostic scores in the wait list group after no treatment at times 1 and 2; Test type: Superiority or Other; p < 0.001, Chi-squared; % of participants with PCL score > 50 = 41.0
Statistical Analysis 3: Comparison: Wait List: Thought Field Therapy; Test type: Superiority or Other; p < 0.001, Chi-squared; Percentage = 39.9

3. Post Hoc Outcome: Assessment of Any Persisting Benefit of TFT (Thought Field Therapy) After 19 Months.
Description: PCL-C (post traumatic check list for civilians) is a measure of the severity of post traumatic stress disorder (PTSD), and can also be used for screening populations, It is a self-completed questionnaire with 17 questions scoring from 1 - 5. The scores of each question are added to create the total score for each participant. The highest possible score for any individual is 85, the lowest score being 17. A diagnostic score for PTSD is accepted as being more than 50. Participants completed the PCL-C one week following treatment and nineteen months later. Comparison of PCL-C scores at nineteen months compared to one week following treatment.
Time Frame: 1 week post-treatment (Time 2, TFT; Time 3, WL) and 19 months later.
Population: All those who had scores one week after treatment and at 19 months. Similar gender and age proportions to original groups.
Measure: Mean (Standard Deviation); unit: units on a scale (PCL-C score)
Arm/Group | Thought Field Therapy
Number analyzed (Participants) | 116
units on a scale (PCL-C score)
  one week following treatment | 25.8 (7.8)
  19 months later | 43.6 (13.1)
Statistical Analysis 1: Comparison: Thought Field Therapy; Both the original treatment and control groups were combined as both groups had been treated at a similar time before the nineteen month assessment. The null hypothesis was that there had been no change in the PCL-C scores at nineteen months compared to one week following treatment; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 17.8, 95% CI 2-sided [15.2 to 20.5]

4. Post Hoc Outcome: Assessment of Continuing Benefit of TFT After 19 Months, in Control Group, as Measured by a Diagnosis of PTSD According to a PCL-C Score of >50.
Description: PCL-C (post traumatic check list for civilians) is a measure of the severity of post traumatic stress disorder (PTSD), and can also be used for screening populations, It is a self-completed questionnaire with 17 questions scoring from 1 - 5. The scores of each question are added to create the total score for each participant. The highest possible score for any individual is 85, the lowest score being 17. A diagnostic score for PTSD is accepted as being more than 50. Participants completed the PCL-C just before treatment and one week later. Only the wait-list control group was used as the treatment group did not not have a run-in score, and would have given inappropriately positive results.
Time Frame: Time 2 and 19 months later.
Population: 83% female average age 43 years, 17% male average age 46.7 years.
Measure: Number; unit: percentage of PCL-C scores >50.
Groups:
- Wait List Group: Those in the wait list, who had attended for their second immediate pre-treatment assessment and attended for assessment 19 months later.
Arm/Group | Wait List Group
Number analyzed (Participants) | 71
percentage of PCL-C scores >50.
  PCL-C score pre-treatment (time 2) >50 | 41.8
  % with PCL-C score >50 at 19 months | 26.6

ADVERSE EVENTS:
Time Frame: Complete up to time 3, that is one week after treatment. Incomplete up to 19 months later.
Description: Adverse events were reported for all those who were treated. There were 128 in the treatment group, but only 122 in the waitlist group as four did not attend for treatment at time 2, making 250 in total.
Groups:
- Thought Field Therapy: Thought Field Therapy delivered by trained community leaders.
  Thought Field Therapy.: Thought Field Therapy is a meridian based therapy, where clients tap on specific parts of their body, according to a particular protocol. This does not obliterate the memory of the trauma, but relieves the associated distress.
  Both groups were invited to attend 19 months later
Arm/Group | Thought Field Therapy
Serious Adverse Events (participants affected / at risk) | 1/250
Other Adverse Events (participants affected / at risk) | 2/250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thought Field Therapy (N=250)
Death (Social circumstances) | 1 (1) — Cause unknown
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thought Field Therapy (N=250)
Functional seizure (Psychiatric disorders) | 1 (1) — Known history of blackouts, likely to be non-organic. One occurred during therapy with complete recovery.
Hysterical reaction (Psychiatric disorders) | 1 (1) — Uncontrollable shaking and rapid speech

LIMITATIONS AND CAVEATS:
Only one assessment tool for PTSD was used. The 19 month data interpretation was limited by the high drop-out rate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No